CLINICAL TRIAL: NCT00004160
Title: Sequential and Concomitant Chemoradiotherapy With Gemcitabine-Based Chemotherapy for Inoperable Stage IIIa and IIIb Non-Small Cell Lung Cancer: A Phase I/IIa Study
Brief Title: Chemotherapy Plus Radiation Therapy in Treating Patients With Stage III Non-small Cell Lung Cancer That Cannot Be Surgically Removed
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067400; UAB-9718; UAB-F97073005; NCI-G99-1625
Record Dates: First submitted 1999-12-10; First posted 2004-07-19 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2005-10

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Gemcitabine; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Dose 1 Gemcitabine (Experimental): Patients receive paclitaxel IV over 1 hour and gemcitabine IV over 30 minutes beginning 2 hours into paclitaxel infusion on day 1 of weeks 6, 9, and 12.
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride; Drug: paclitaxel; Radiation: radiation therapy
- Dose 2 Gemcitabine (Experimental): Patients receive paclitaxel IV over 1 hour and gemcitabine IV over 30 minutes beginning 2 hours into paclitaxel infusion on day 1 of weeks 6, 9, and 12.
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride; Drug: paclitaxel; Radiation: radiation therapy
- Dose 3 Gemcitabine (Experimental): Patients receive paclitaxel IV over 1 hour and gemcitabine IV over 30 minutes beginning 2 hours into paclitaxel infusion on day 1 of weeks 6, 9, and 12.
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride; Drug: paclitaxel; Radiation: radiation therapy
- Dose 4 Gemcitabine (Experimental): Patients receive paclitaxel IV over 1 hour and gemcitabine IV over 30 minutes beginning 2 hours into paclitaxel infusion on day 1 of weeks 6, 9, and 12.
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride; Drug: paclitaxel; Radiation: radiation therapy
- Dose 5 Gemcitabine (Experimental): Patients receive paclitaxel IV over 1 hour and gemcitabine IV over 30 minutes beginning 2 hours into paclitaxel infusion on day 1 of weeks 6, 9, and 12.
  Interventions: Drug: cisplatin; Drug: gemcitabine hydrochloride; Drug: paclitaxel; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of chemotherapy plus radiation therapy in treating patients who have stage III non-small cell lung cancer that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and dose limiting toxicity of gemcitabine and paclitaxel in combination with radiotherapy in patients with locally advanced stage IIIA or IIIB non-small cell lung cancer. II. Assess response rate, duration of response, disease free survival and failure in this patient population on this regimen. III. Determine the pharmacokinetics of gemcitabine and paclitaxel during the chemoradiotherapy phase.

OUTLINE: This is a dose escalation study of gemcitabine. Induction phase: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and cisplatin IV over 1 hour on day 1. Treatment repeats every 3 weeks for 2 courses. Chemoradiotherapy phase: Patients receive paclitaxel IV over 1 hour and gemcitabine IV over 30 minutes beginning 2 hours into paclitaxel infusion on day 1 of weeks 6, 9, and 12. Patients undergo conventional chest radiotherapy on Monday though Friday for weeks 6-11. Cohorts of 3-5 patients receive escalating doses of gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which at least 2 of 5 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: A minimum of 17 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed locally advanced, unresectable non- small cell lung cancer Stage IIIA or IIIB Local, unresectable recurrence after primary surgery allowed Measurable or evaluable disease No contralateral pleural effusion(s) or noncontiguous pleural implants T4 tumors with small ipsilateral pleural effusions allowed

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT or SGPT no greater than 2 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No prior myocardial infarction within the past 6 months No congestive heart failure No uncontrolled arrhythmias Pulmonary: FEV1 greater than 800 mL Other: Not pregnant Negative pregnancy test Fertile patients must use effective contraception No history of hypersensitivity to drugs formulated in Cremophor EL No other malignancy within the past 5 years, except: Nonmelanomatous skin cancer Carcinoma in situ of the cervix No overt psychosis or other major debilitating disorder that would preclude compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2000-02; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose and dose limiting toxicity of gemcitabine and paclitaxel in combination with radiotherapy in patients with locally advanced stage IIIA or IIIB non-small cell lung cancer. | baseline to 6 - 11 weeks

SECONDARY OUTCOMES:
Assess response rate, duration of response, disease free survival and failure in this patient population on this regimen. | baseline to 6 - 11 weeks
Determine the pharmacokinetics of gemcitabine and paclitaxel during the chemoradiotherapy phase | baseline to 6 - 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, MD, FACP, Study Chair — University of Alabama at Birmingham
Locations (1):
- University of Alabama Comprehensive Cancer Center, Birmingham, Alabama, United States

REFERENCES:
- [Result] Divers SG, Spencer SA, Carey D, Busby EM, Hyatt MD, Robert F. Phase I/IIa study of cisplatin and gemcitabine as induction chemotherapy followed by concurrent chemoradiotherapy with gemcitabine and paclitaxel for locally advanced non-small-cell lung cancer. J Clin Oncol. 2005 Sep 20;23(27):6664-73. doi: 10.1200/JCO.2005.02.519. PMID 16170174